CLINICAL TRIAL: NCT05484310
Title: Randomized Multicenter Comparison Between Ultrathin-strut Biodegradable Polymer Sirolimuseluting Stents and Durable Polymer Everolimus-eluting Stents for Patients With Acute ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: BIOSTEMI Extended Survival
Acronym: BIOSTEMI ES
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, IGLESIAS Juan Fernando, PD Dr, University Hospital, Geneva
Other Study IDs: 2021-01928
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: ST-segment elevation myocardial infarction; Long-term outcomes; Primary PCI
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the BIOSTEMI ES study is to assess the long-term clinical outcomes with the Orsiro ultrathin-strut biodegradable polymer sirolimus-eluting stent compared to the Xience thin-strut durable polymer everolimus-eluting stent up to 5 years of follow-up among patients with STEMI undergoing primary PCI, enrolled in the BIOSTEMI trial.

DETAILED DESCRIPTION:
The objective of the BIOSTEMI ES study is to assess the long-term clinical outcomes with the Orsiro ultrathin-strut biodegradable polymer sirolimus-eluting stent compared to the Xience thin-strut durable polymer everolimus-eluting stent up to 5 years of follow-up among patients with STEMI undergoing primary PCI, enrolled in the BIOSTEMI trial.

* In the BIOSTEMI randomized controlled clinical trial, the Orsiro ultrathin-strut bio degradable polymer sirolimus-eluting stent was found superior to the best-in-class Xience thin-strut durable polymer everolimus-eluting stent with respect to target lesion failure at one-year follow-up among patients with STEMI undergoing primary PCI (Iglesias JF, et al., Lancet 2019). The difference was driven by a lower risk of clinically indicated target lesion revascularization with the Orsiro ultrathin-strut biodegradable polymer sirolimus-eluting stent compared to the Xience thin-strut durable polymer everolimus-eluting stent.
* Importantly, the difference between Orsiro stent and Xience stent accrues over time between one and two years of follow-up.
* As per study protocol, the planned follow-up of patients included in the BIOSTEMI randomized controlled trial was 2 years.
* The long-term clinical benefits the Orsiro ultrathin-strut biodegradable polymer sirolimus-eluting stent over the Xience thin-strut durable polymer everolimus-eluting stent beyond the polymer degradation period remain uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that were enrolled in the BIOSTEMI trial (BASEC: 2016-00555),
* Subject willing and able to provide oral informed consent.

Exclusion Criteria:

* No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BIOSTEMI ES includes only participants of the BIOSTEMI trial, i.e. patients with acute STEMI presenting within 24 hours of symptom onset undergoing primary PCI. At PCI, the randomly allocated stent (Orsiro® vs Xience®) was implanted in the culprit lesion of the target vessel.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Target lesion failure, composite of cardiac death, target vessel (Q-wave or non-Q-wave) myocardial re-infarction, or clinically indicated target lesion revascularization | 5 years of follow-up
  Clinical assessment

SECONDARY OUTCOMES:
Cardiac death | 5 years of follow-up
  Clinical assessment
All-cause death | 5 years of follow-up
  Clinical assessment
Target vessel myocardial re-infarction | 5 years of follow-up
  Clinical assessment
Any myocardial infarction (Q-wave and non-Q-wave) | 5 years of follow-up
  Clinical assessment
Clinically indicated and not clinically indicated target lesion revascularization | 5 years of follow-up
  Clinical assessment
Clinically indicated and not clinically indicated target vessel revascularization | 5 years of follow-up
  Clinical assessment
Any revascularization | 5 years of follow-up
  Clinical assessment
Target vessel failure, composite of cardiac death, target vessel myocardial re-infarction, or clinically indicated target vessel revascularization | 5 years of follow-up
  Clinical assessment
Definite stent thrombosis | 5 years of follow-up
  Clinical assessment
Definite/probable stent thrombosis | 5 years of follow-up
  Clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Pr, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Juan F. Iglesias, PD Dr, Principal Investigator — University Hospital, Geneva
Locations (10):
- Switzerland (10):
  - Kantonsspital Aarau, Aarau
  - Basel University Hospital, Basel
  - Inselspital, Bern University Hospital, Bern
  - Hôpital Cantonal de Fribourg, Fribourg
  - Geneva University Hospitals, Geneva
  - Lausanne University Hospitals, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St.Gallen, Sankt Gallen
  - Spital Wallis, Sion
  - Triemli Hospital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan will depend on editorial publication policies requirements.

REFERENCES:
- [Background] Iglesias JF, Muller O, Zaugg S, Roffi M, Kurz DJ, Vuilliomenet A, Weilenmann D, Kaiser C, Tapponnier M, Heg D, Valgimigli M, Eeckhout E, Juni P, Windecker S, Pilgrim T. A comparison of an ultrathin-strut biodegradable polymer sirolimus-eluting stent with a durable polymer everolimus-eluting stent for patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: rationale and design of the BIOSTEMI trial. EuroIntervention. 2018 Aug 20;14(6):692-699. doi: 10.4244/EIJ-D-17-00734. PMID 29205157
- [Background] Iglesias JF, Muller O, Heg D, Roffi M, Kurz DJ, Moarof I, Weilenmann D, Kaiser C, Tapponnier M, Stortecky S, Losdat S, Eeckhout E, Valgimigli M, Odutayo A, Zwahlen M, Juni P, Windecker S, Pilgrim T. Biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents in patients with ST-segment elevation myocardial infarction (BIOSTEMI): a single-blind, prospective, randomised superiority trial. Lancet. 2019 Oct 5;394(10205):1243-1253. doi: 10.1016/S0140-6736(19)31877-X. Epub 2019 Sep 2. PMID 31488372
- [Background] Pilgrim T, Muller O, Heg D, Roffi M, Kurz DJ, Moarof I, Weilenmann D, Kaiser C, Tapponnier M, Losdat S, Eeckhout E, Valgimigli M, Juni P, Windecker S, Iglesias JF. Biodegradable- Versus Durable-Polymer Drug-Eluting Stents for STEMI: Final 2-Year Outcomes of the BIOSTEMI Trial. JACC Cardiovasc Interv. 2021 Mar 22;14(6):639-648. doi: 10.1016/j.jcin.2020.12.011. PMID 33727005
- [Derived] Iglesias JF, Roffi M, Losdat S, Muller O, Degrauwe S, Kurz DJ, Haegeli L, Weilenmann D, Kaiser C, Tapponnier M, Cook S, Cuculi F, Heg D, Windecker S, Pilgrim T. Long-term outcomes with biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents in ST-segment elevation myocardial infarction: 5-year follow-up of the BIOSTEMI randomised superiority trial. Lancet. 2023 Nov 25;402(10416):1979-1990. doi: 10.1016/S0140-6736(23)02197-9. Epub 2023 Oct 25. PMID 37898137